CLINICAL TRIAL: NCT03596424
Title: Impact of Dexmedetomidine and Ketamine and Their Combination for the Reduction of Postoperative Morphine Requirements After VATS Surgery
Brief Title: Dexmedetomidine and Ketamine in VATS Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Dr, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DexketVATS
Record Dates: First submitted 2018-05-27; First posted 2018-07-23 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine hydrochloride (Active Comparator): Intraoperative bolus (0.25 mg/kg) and infusion (0.25mg/kg/h) of ketamine plus an intraoperative bolus (over 20 min) and infusion of normal saline;
  Interventions: Drug: Ketamine Hydrochloride
- dexmedetomidine hydrochloride (Active Comparator): Intraoperative bolus (1µg/kg over 20 min) and infusion (0.5µg/kg/h) of dexmedetomidine plus an intraoperative bolus and infusion of normal saline
  Interventions: Drug: Dexmedetomidine Hydrochloride
- dexmedetomidine hydrochloride and ketamine hydrochloride (Active Comparator): Intraoperative bolus (1µg/kg over 20 min) and infusion (0.5 µg/g/h) of dexmedetomidine plus an intraoperative bolus (0.25mg/kg) and infusion (0.25mg/kg/h) of ketamine
  Interventions: Combination Product: dexmedetomidine Hydrochloride and Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Intraoperative bolus and infusion (see arm description)
  Other Names: ketamine
  Arms: Ketamine hydrochloride
Drug: Dexmedetomidine Hydrochloride — Intraoperative bolus and infusion (see arm description)
  Other Names: dexmedetomidine
  Arms: dexmedetomidine hydrochloride
Combination Product: dexmedetomidine Hydrochloride and Ketamine Hydrochloride — Intraoperative bolus and infusion (see arm description)
  Other Names: dexmedetomidine and ketamine
  Arms: dexmedetomidine hydrochloride and ketamine hydrochloride

SUMMARY:
Postoperative pain after VATS surgery is significant and associated with moderate to high post operative morphine requirements, which can cause opioid related side effects and delay postoperative recovery. To reduce this requirement, multimodal analgesia with non opioid medication such as dexmedetomidine and ketamine can be used. These drugs have demonstrated significant opioid-sparing properties after various types of surgeries. However, very little is known about their ability to do so in VATS surgery. Also, their relative opioid-sparing properties have not been compared, and it is not known whether their combined use can lead to an additional opioid-sparing effect. The primary goal of this study will be to determine the impact of a combined intra operative infusion of ketamine and dexmedetomidine on postoperative morphine requirements in patients undergoing elective VATS, compared to both these drugs infused separately.

The hypothesis is that this combined infusion will lead to a 30% further reduction in morphine requirements, 24h after surgery, compared to both these drugs infused separately.

DETAILED DESCRIPTION:
Video-assisted thoracic surgery (VATS) for pulmonary resection is associated with less tissue trauma, less impairment in lung function, and reduced postoperative pain compared with thoracotomy, although many patients continue to report significant acute postoperative pain. If not well-controlled, postoperative thoracic pain can lead to splinting and inadequate recovery of pulmonary function.

Enhancing the quality of postoperative analgesia while reducing intra and postoperative opioid requirements is an important issue that has been one of the main focus of Enhanced Recovery After Surgery (ERAS) protocols. Indeed, the key factors that delay postoperative recovery include parenteral opioids and bed rest and immobility secondary to postoperative pain. While opioids are effective at treating even severe pain, their use is associated with dose-related adverse effects such as respiratory depression, sedation, postoperative nausea and vomiting, urinary retention, ileus, opioid-induced hyperalgesia and chronic postoperative pain. More importantly, opioids depress host immunity and neuroendocrine function and may negatively affect cancer recurrence and survival after lung cancer surgery.

Hence, given the importance of good postoperative analgesia and the significance of opioid-related adverse effects, the reduction of opioid requirements and postoperative pain through multimodal analgesia is an important matter. Focusing on this goal, the ERAS protocols have shown great efficacy in improving patient's care after colorectal surgery and they are now being applied to pancreatic, ENT, bariatric, urologic and many more major surgeries.

It is probably only a matter of time before ERAS protocols are applied to VATS surgery; however, the optimal way of providing postoperative analgesia after VATS has not yet been determined, unlike colorectal surgery. Indeed, thoracic epidural analgesia, single-shot and continuous paravertebral and intercostal nerve blocks and patient-controlled intravenous analgesia have all been evaluated, and none of these has consistently emerged as being superior to the others or to intravenous analgesia. Thoracic epidural analgesia provides effective pain control for thoracotomy but its benefits following thoracoscopy are not uniform. Furthermore, the risks of sympathectomy-induced hypotension and neurologic injury from epidural hematoma may not be justified considering the lesser postoperative pain and impairment in pulmonary function compared to thoracotomy. Continuous paravertebral blocks are an effective alternative to epidural analgesia although their performance may be challenging and time consuming, and catheters may be difficult to thread or get accidentally removed, leading to block failure. Furthermore, as for epidural analgesia, paravertebral catheter placement is contra-indicated in patients with impaired coagulation and/or infection. Single-shot intercostal and paravertebral blocks are less invasive although their benefit is restricted to the first twelve postoperative hours.

Moreover, none of these regional anesthesia techniques can treat the ipsilateral shoulder pain that is often associated with VATS, and opioid analgesia might still be required.

An intravenous opioid patient-controlled analgesia combined to multimodal analgesia with acetaminophen and non-steroidal anti-inflammatoy drug (NSAID) is commonly used in many institutions and has shown to provide adequate and effective postoperative analgesia. However, significant acute postoperative pain and moderate to high opioid consumption are still reported after VATS. There is definitely some place for improvement, which could come from other non-opioid analgesic adjuncts such as ketamine and/or dexmedetomidine.

Ketamine is an anesthetic drug that has well-known analgesic properties due to its ability to block NMDA receptors. An intraoperative bolus followed with a low-dose infusion reduces postoperative opioid requirements by 30-40%, without causing significant side effects. Similarly, dexmedetomidine is a centrally acting α2-agonist with sedating and analgesic properties. When used intra-operatively, it significantly reduces hypnotics and opioids requirements, decreases median pain scores and reduces postoperative morphine consumption by approximately 30%. These systematic reviews seem to indicate a greater morphine-sparing effect from ketamine compared to dexmedetomidine although this has not been evaluated thoroughly. Indeed, only one study compared ketamine's morphine-sparing effects to that of dexmedetomidine, in patients undergoing spine surgery. Both infusions were started postoperatively and provided significant morphine sparing effects compared to placebo. Ketamine's morphine-sparing effect appeared greater than that of dexmedetomidine, although this was not statistically significant, as this study was not powered for that outcome. Hence, their morphine-sparing effect might be different but this difference is likely small. Their impact on postoperative opioid requirement after VATS surgery has not been studied, even though it could be highly beneficial, not only for the reduction of postoperative opioid requirements but for the reduction of chronic postoperative pain.

Another interesting reason for using these analgesic adjuvants for intra operative analgesia is their ability to prevent chronic post operative pain.

More interesting would be to investigate whether their combined use leads to greater morphine-sparing effect. Indeed, although their combination for paediatric procedural sedation is well described, the impact of a combined dexmedetomidine-ketamine intraoperative infusion on postoperative analgesia and opioid requirements has not been evaluated.

Study outcome and hypothesis

The primary goal of this study will be to determine the impact of a combined intra operative infusion of ketamine and dexmedetomidine on postoperative morphine requirements in patients undergoing elective VATS, compared to both these drugs infused separately.

The hypothesis is that this combined infusion will lead to a 30% further reduction in morphine requirements, 24h after surgery, compared to both these drugs infused separately.

Secondary outcomes will be to evaluate the impact of a combined dexmedetomidine-ketamine infusion on:

* Postoperative pain scores at rest and after coughing at 24 and 48 h postoperatively;
* Cumulative morphine consumption 48 h after surgery;
* Intraoperative fentanyl requirements, determined using the NoL index (see methodology section, page);
* Time to chest tube removal and time to hospital discharge;
* Proportion of patients with persistent pain three months after surgery;
* Incidence of ketamine-induced psychomimetic side effects in the postoperative period
* Incidence of intraoperative bradycardia <50 beats/min compared to intraoperative infusions of ketamine only and dexmedetomidine only.

METHODOLOGY

Study design

This will be a prospective, randomized, double blind study.

Population

Patients undergoing elective VATS and receiving an opioid intravenous patient-controlled analgesia (PCA) combined with acetaminophen and NSAID for postoperative analgesia.

Duration of study

1 year

Sample size Postoperative cumulative morphine consumption 24h after surgery in our institution has been determined by reviewing the files of 50 patients who underwent VATS surgery and received a PCA combined to acetaminophen and NSAID for postoperative analgesia. These patients used an average (standard deviation (SD)) of 39.5 (17.3) mg of morphine.

Considering an opioid-sparing effect of 30% from dexmedetomidine and ketamine alone, a mean morphine consumption of 27.7(11) mg can be expected in the ketamine and dexmedetomidine groups.

A 30% further reduction in opioid requirement from combining ketamine to dexmedetomidine will be considered significant.

Thus, a sample size of 37 patients per group would give us 80% power to detect such a difference, alpha 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old
* American Society of Anesthesiology physical status I-III
* Elective Video-Assisted Thoracic Surgery for pulmonary resection

Exclusion Criteria:

* Patients for which a regional anesthesia technique is planned for postoperative analgesia.
* Patients taking beta-blockers preoperatively.
* Patients with chronic pain taking >60 mg morphine PO daily (or its equivalent).
* Patients taking pregabalin, gabapentin, amitryptillin, nortryptillin and/or duloxetin.
* Documented allergy to ketamine and/or dexmedetomidine.
* Pregnancy
* Inability to give informed consent
* Linguistic barrier.
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Day 1 Postoperative morphine requirement | Day 1
  Cumulative dose of morphine used by the patient

SECONDARY OUTCOMES:
day 2 Postoperativve morphine requirement | day 2
  cumulative dose of morphine used by the patient
Pain score at rest 24h | day 1
  Pain score (Verbal Numeric Scale (0-10) at rest
Pain score at rest 48h | day 2
  Pain score (Verbal Numeric Scale (0-10) at rest
Pain score at cough 24h | day 1
  Pain score (Verbal Numeric Scale (0-10) at cough
Pain score at cough 48h | day 2
  Pain score (Verbal Numeric Scale (0-10) at cough
intraoperative fentanyl requirement | for incision to wound closure
  intraoperative dose of fentanyl used to treat intraoperative pain
chest tube removal | 1 week
  time (days) for chest tube removal after surgery
chronic postoperative pain | 3 months
  patients reporting persistent post operative pain

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Ciusss, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No